CLINICAL TRIAL: NCT01601223
Title: Local Assessment of Ventilatory Management During General Anesthesia for Surgery - a Prospective Observational Multi-center Cohort Study
Brief Title: Local Assessment of Ventilatory Management During General Anesthesia for Surgery
Acronym: LAS VEGAS
Status: Completed | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Other Study IDs: LAS VEGAS
Record Dates: First submitted 2012-05-14; First posted 2012-05-17 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Surgery; Anaesthesia; Ventilator-Induced Lung Injury; Lung Injury; Pneumonia; Pneumothorax; Respiratory Distress Syndrome, Adult; Respiratory Insufficiency
Keywords: Ventilatory Management; Mechanical Ventilation; Post Operative pulmonary complications; Intra-operative complications; General Anesthesia; Surgery; LAS VEGAS; ESA (European Society of Anaesthesiology); European Society of Anaesthesiology
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Lung Injury; Pneumonia; Pneumothorax; Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical mechanically-ventilated: Surgical patients undergoing invasive mechanical ventilation for general anesthesia

SUMMARY:
Objectives

1. To characterize mechanical ventilation practices during general anesthesia for surgery
2. To assess the dependence of intra-operative and post-operative pulmonary complications on intra-operative Mechanical Ventilation (MV) settings

DETAILED DESCRIPTION:
Research questions

* What MV-settings are used during general anesthesia for surgery?
* Do MV-settings vary in and/or between centers?
* Do MV-settings vary internationally?
* Are MV-settings associated with incidence of intra-operative pulmonary complications?
* Are MV-settings associated with incidence of post-operative pulmonary complications?

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* All surgical procedures requiring invasive mechanical ventilation (MV)during general anesthesia for laparoscopic or non-laparoscopic surgery.
* This includes MV performed with supra-glottic devices (e.g. laryngeal mask)
* This includes patients receiving MV at the onset of the procedure (e.g. Intensive Care Unit patients)
* This includes patients who will receive one-lung ventilation during the procedure

Exclusion Criteria:

* Obstetric surgical procedures or any procedure during pregnancy
* Surgical procedures outside the operating room
* Surgical procedures involving extra-corporal circulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients undergoing general anesthesia for surgery during a period of one week
Sampling Method: Non-Probability Sample
Enrollment: 10690 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Post-operative pulmonary complications, possibly related to ventilation strategy | Post-operative on day of surgery, day 1, 2,3,4,5 and day 28
  Effect of Mechanical Ventilation settings during general anesthesia for surgery on the incidence of post-operative pulmonary complications (new or prolonged invasive or non-invasive mechanical ventilation, need for oxygen therapy, respiratory failure, pneumonia, ARDS 'Acute Respiratory Distress Syndrome', pneumothorax) Defined post-operative pulmonary complications are recorded from the medical chart on day 0, 1, 2, 3, 4 and 5 after surgery. On day 28 length of hospital stay and in hospital death are assessed.

SECONDARY OUTCOMES:
Intra-operative complications related to the ventilation strategy | Time point(s) at which outcome measure is assessed is is: Day of surgery, day 1, 2, 3, 4, 5 and 28 after surgery
Mechanical ventilation-settings during general anesthesia for surgery | During the surgical procedure, from moment of to tracheal extubation or discharge from operation room (in case patient remains on mechanical ventilation)
  * Variation of applied MV settings within centers
  * Variation of applied MV settings between centers on an international basis

CONTACTS AND LOCATIONS:
Overall Officials: Schultz Marcus, MD, Study Chair — AMC, Amsterdam, The Netherlands; Sabrine Hemmes, MD, Study Director — AMC, Amsterdam, The Netherlands
Locations (19):
- United States (3):
  - University of Colorado School of Medicine/University of Colorado Hospital, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
- Estonia (2):
  - North Estonia Medical Center, Tallinn
  - Tartu University Hospital, Tartu
- Germany (3):
  - University Hospital Carl Gustav Carus, Dresden University of Technonology, Department of Anesthesiology and Intensive Care Therapy, Dresden
  - Duesseldorf University Hospital, Düsseldorf
  - Diakoniekrankenhaus Friederikenstift, Hanover
- Italy (2):
  - Ospedale San Martino, Dipartimento di scienze chirurgiche e diagnostiche integrate, Genoa
  - Ospedale San Raffaele, Milan
- Lithuania (2):
  - Vilnius University Hospital - Institute of Oncology, Vilnius
  - Vilnius University Hospital - Santariskiu Clinics, Vilnius
- Netherlands (3):
  - Academic Medical Center, University of Amsterdam, Amsterdam
  - VU University Medical Center, Amsterdam
  - MC Haaglanden, The Hague
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Førde Central Hospital /Førde Sentral Sykehus, Førde
- Slovenia (2):
  - Institute of Oncology Ljubljana, Ljubljana
  - University Medicine Centre Ljubljana, Ljubljana

REFERENCES:
- [Background] Putensen C, Theuerkauf N, Zinserling J, Wrigge H, Pelosi P. Meta-analysis: ventilation strategies and outcomes of the acute respiratory distress syndrome and acute lung injury. Ann Intern Med. 2009 Oct 20;151(8):566-76. doi: 10.7326/0003-4819-151-8-200910200-00011. PMID 19841457
- [Background] Tremblay LN, Slutsky AS. Ventilator-induced lung injury: from the bench to the bedside. Intensive Care Med. 2006 Jan;32(1):24-33. doi: 10.1007/s00134-005-2817-8. Epub 2005 Oct 18. No abstract available. PMID 16231069
- [Background] Slutsky AS. Lung injury caused by mechanical ventilation. Chest. 1999 Jul;116(1 Suppl):9S-15S. doi: 10.1378/chest.116.suppl_1.9s-a. No abstract available. PMID 10424561
- [Background] Burns KE, Adhikari NK, Slutsky AS, Guyatt GH, Villar J, Zhang H, Zhou Q, Cook DJ, Stewart TE, Meade MO. Pressure and volume limited ventilation for the ventilatory management of patients with acute lung injury: a systematic review and meta-analysis. PLoS One. 2011 Jan 28;6(1):e14623. doi: 10.1371/journal.pone.0014623. PMID 21298026
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Gajic O, Frutos-Vivar F, Esteban A, Hubmayr RD, Anzueto A. Ventilator settings as a risk factor for acute respiratory distress syndrome in mechanically ventilated patients. Intensive Care Med. 2005 Jul;31(7):922-6. doi: 10.1007/s00134-005-2625-1. Epub 2005 Apr 26. PMID 15856172
- [Background] Gajic O, Dara SI, Mendez JL, Adesanya AO, Festic E, Caples SM, Rana R, St Sauver JL, Lymp JF, Afessa B, Hubmayr RD. Ventilator-associated lung injury in patients without acute lung injury at the onset of mechanical ventilation. Crit Care Med. 2004 Sep;32(9):1817-24. doi: 10.1097/01.ccm.0000133019.52531.30. PMID 15343007
- [Background] Briel M, Meade M, Mercat A, Brower RG, Talmor D, Walter SD, Slutsky AS, Pullenayegum E, Zhou Q, Cook D, Brochard L, Richard JC, Lamontagne F, Bhatnagar N, Stewart TE, Guyatt G. Higher vs lower positive end-expiratory pressure in patients with acute lung injury and acute respiratory distress syndrome: systematic review and meta-analysis. JAMA. 2010 Mar 3;303(9):865-73. doi: 10.1001/jama.2010.218. PMID 20197533
- [Background] Lachmann B. Open up the lung and keep the lung open. Intensive Care Med. 1992;18(6):319-21. doi: 10.1007/BF01694358. No abstract available. PMID 1469157
- [Background] Fernandez-Perez ER, Keegan MT, Brown DR, Hubmayr RD, Gajic O. Intraoperative tidal volume as a risk factor for respiratory failure after pneumonectomy. Anesthesiology. 2006 Jul;105(1):14-8. doi: 10.1097/00000542-200607000-00007. PMID 16809989
- [Background] Schultz MJ, Haitsma JJ, Slutsky AS, Gajic O. What tidal volumes should be used in patients without acute lung injury? Anesthesiology. 2007 Jun;106(6):1226-31. doi: 10.1097/01.anes.0000267607.25011.e8. PMID 17525599
- [Background] Wrigge H, Uhlig U, Baumgarten G, Menzenbach J, Zinserling J, Ernst M, Dromann D, Welz A, Uhlig S, Putensen C. Mechanical ventilation strategies and inflammatory responses to cardiac surgery: a prospective randomized clinical trial. Intensive Care Med. 2005 Oct;31(10):1379-87. doi: 10.1007/s00134-005-2767-1. Epub 2005 Aug 17. PMID 16132888
- [Background] Wrigge H, Uhlig U, Zinserling J, Behrends-Callsen E, Ottersbach G, Fischer M, Uhlig S, Putensen C. The effects of different ventilatory settings on pulmonary and systemic inflammatory responses during major surgery. Anesth Analg. 2004 Mar;98(3):775-81, table of contents. doi: 10.1213/01.ane.0000100663.11852.bf. PMID 14980936
- [Background] Wolthuis EK, Choi G, Dessing MC, Bresser P, Lutter R, Dzoljic M, van der Poll T, Vroom MB, Hollmann M, Schultz MJ. Mechanical ventilation with lower tidal volumes and positive end-expiratory pressure prevents pulmonary inflammation in patients without preexisting lung injury. Anesthesiology. 2008 Jan;108(1):46-54. doi: 10.1097/01.anes.0000296068.80921.10. PMID 18156881
- [Background] Rothen HU, Sporre B, Engberg G, Wegenius G, Reber A, Hedenstierna G. Prevention of atelectasis during general anaesthesia. Lancet. 1995 Jun 3;345(8962):1387-91. doi: 10.1016/s0140-6736(95)92595-3. PMID 7760608
- [Background] Blum JM, Maile M, Park PK, Morris M, Jewell E, Dechert R, Rosenberg AL. A description of intraoperative ventilator management in patients with acute lung injury and the use of lung protective ventilation strategies. Anesthesiology. 2011 Jul;115(1):75-82. doi: 10.1097/ALN.0b013e31821a8d63. PMID 21552117
- [Background] Schultz MJ. Lung-protective mechanical ventilation with lower tidal volumes in patients not suffering from acute lung injury: a review of clinical studies. Med Sci Monit. 2008 Feb;14(2):RA22-26. PMID 18227773
- [Background] Imberger G, McIlroy D, Pace NL, Wetterslev J, Brok J, Moller AM. Positive end-expiratory pressure (PEEP) during anaesthesia for the prevention of mortality and postoperative pulmonary complications. Cochrane Database Syst Rev. 2010 Sep 8;(9):CD007922. doi: 10.1002/14651858.CD007922.pub2. PMID 20824871
- [Background] Tusman G, Bohm SH. Prevention and reversal of lung collapse during the intra-operative period. Best Pract Res Clin Anaesthesiol. 2010 Jun;24(2):183-97. doi: 10.1016/j.bpa.2010.02.006. PMID 20608556
- [Background] Smetana GW, Lawrence VA, Cornell JE; American College of Physicians. Preoperative pulmonary risk stratification for noncardiothoracic surgery: systematic review for the American College of Physicians. Ann Intern Med. 2006 Apr 18;144(8):581-95. doi: 10.7326/0003-4819-144-8-200604180-00009. PMID 16618956
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Bagley SC, White H, Golomb BA. Logistic regression in the medical literature: standards for use and reporting, with particular attention to one medical domain. J Clin Epidemiol. 2001 Oct;54(10):979-85. doi: 10.1016/s0895-4356(01)00372-9. PMID 11576808
- [Background] Winkel TA, Schouten O, Hoeks SE, Flu WJ, Hampton D, Kirchhof P, van Kuijk JP, Lindemans J, Verhagen HJ, Bax JJ, Poldermans D. Risk factors and outcome of new-onset cardiac arrhythmias in vascular surgery patients. Am Heart J. 2010 Jun;159(6):1108-15. doi: 10.1016/j.ahj.2010.03.035. PMID 20569727
- [Background] Murphy GS, Brull SJ. Residual neuromuscular block: lessons unlearned. Part I: definitions, incidence, and adverse physiologic effects of residual neuromuscular block. Anesth Analg. 2010 Jul;111(1):120-8. doi: 10.1213/ANE.0b013e3181da832d. Epub 2010 May 4. PMID 20442260
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Background] Hemmes SN, de Abreu MG, Pelosi P, Schultz MJ. ESA Clinical Trials Network 2012: LAS VEGAS--Local Assessment of Ventilatory Management during General Anaesthesia for Surgery and its effects on Postoperative Pulmonary Complications: a prospective, observational, international, multicentre cohort study. Eur J Anaesthesiol. 2013 May;30(5):205-7. doi: 10.1097/EJA.0b013e32835fcab3. No abstract available. PMID 23571432
- [Derived] Dorland G, Saadat W, van Meenen DMP, Neto AS, Hiesmayr M, Hollmann MW, Mills GH, Vidal Melo MF, Putensen C, Schmid W, Severgnini P, Wrigge H, de Abreu MG, Schultz MJ, Hemmes SNT; LAS VEGAS-investigators. Association of preoperative smoking with the occurrence of postoperative pulmonary complications: A post hoc analysis of an observational study in 29 countries. J Clin Anesth. 2025 Jun;104:111856. doi: 10.1016/j.jclinane.2025.111856. Epub 2025 May 14. PMID 40373497
- [Derived] Nasa P, van Meenen DMP, Paulus F, de Abreu MG, Bossers SM, Schober P, Schultz MJ, Neto AS, Hemmes SNT; LAS VEGAS-investigators; PROVE Network; ESAIC CTN; LAS VEGAS collaborators. Associations of intraoperative end-tidal CO2 levels with postoperative outcome-secondary analysis of a worldwide observational study. J Clin Anesth. 2025 Feb;101:111728. doi: 10.1016/j.jclinane.2024.111728. Epub 2024 Dec 19. PMID 39705739
- [Derived] Vermeulen TD, Hol L, Swart P, Hiesmayr M, Mills GH, Putensen C, Schmid W, Serpa Neto A, Severgnini P, Vidal Melo MF, Wrigge H, Hollmann MW, Gama de Abreu M, Schultz MJ, Hemmes SN, van Meenen DM; LAS VEGAS Collaborators group; PROVEnet; Clinical Trial Network of the European Society of Anaesthesiology. Sex dependence of postoperative pulmonary complications - A post hoc unmatched and matched analysis of LAS VEGAS. J Clin Anesth. 2024 Dec;99:111565. doi: 10.1016/j.jclinane.2024.111565. Epub 2024 Sep 23. PMID 39316931
- [Derived] Serafini SC, Hemmes SNT, Serpa Neto A, Schultz MJ, Tschernko E, Gama de Abreu M, Mazzinari G, Ball L; LAS VEGAS - and the AVATaR - investigators. Risk factors for PPCs in laparoscopic non-robotic vs. laparoscopic robotic abdominal surgery (LapRas): rationale and protocol for a patient-level analysis of LAS VEGAS and AVATaR. Rev Esp Anestesiol Reanim (Engl Ed). 2024 Oct;71(8):592-600. doi: 10.1016/j.redare.2024.07.001. Epub 2024 Jul 8. PMID 38987020
- [Derived] Hol L, Nijbroek SGLH, Neto AS, Hemmes SNT, Hedenstierna G, Hiesmayr M, Hollmann MW, Mills GH, Vidal Melo MF, Putensen C, Schmid W, Severgnini P, Wrigge H, de Abreu MG, Pelosi P, Schultz MJ; LAS VEGAS study-investigators. Geo-economic variations in epidemiology, ventilation management and outcome of patients receiving intraoperative ventilation during general anesthesia- posthoc analysis of an observational study in 29 countries. BMC Anesthesiol. 2022 Jan 7;22(1):15. doi: 10.1186/s12871-021-01560-x. PMID 34996361
- [Derived] Mazzinari G, Serpa Neto A, Hemmes SNT, Hedenstierna G, Jaber S, Hiesmayr M, Hollmann MW, Mills GH, Vidal Melo MF, Pearse RM, Putensen C, Schmid W, Severgnini P, Wrigge H, Cambronero OD, Ball L, de Abreu MG, Pelosi P, Schultz MJ; LAS VEGAS study-investigators; PROtective VEntilation NETwork; Clinical Trial Network of the European Society of Anaesthesiology. The Association of Intraoperative driving pressure with postoperative pulmonary complications in open versus closed abdominal surgery patients - a posthoc propensity score-weighted cohort analysis of the LAS VEGAS study. BMC Anesthesiol. 2021 Mar 19;21(1):84. doi: 10.1186/s12871-021-01268-y. PMID 33740885
- [Derived] Nijbroek SG, Hol L, Swart P, Hemmes SNT, Serpa Neto A, Binnekade JM, Hedenstierna G, Jaber S, Hiesmayr M, Hollmann MW, Mills GH, Vidal Melo MF, Putensen C, Schmid W, Severgnini P, Wrigge H, Gama de Abreu M, Pelosi P, Schultz MJ; LAS VEGAS study investigators, the PROVE Network and the Clinical Trial Network of the European Society of Anaesthesiology. Sex difference and intra-operative tidal volume: Insights from the LAS VEGAS study. Eur J Anaesthesiol. 2021 Oct 1;38(10):1034-1041. doi: 10.1097/EJA.0000000000001476. PMID 33606418
- [Derived] Bulte CSE, Boer C, Hemmes SNT, Serpa Neto A, Binnekade JM, Hedenstierna G, Jaber S, Hiesmayr M, Hollmann MW, Mills GH, Vidal Melo MF, Pearse RM, Putensen C, Schmid W, Severgnini P, Wrigge H, Gama de Abreu M, Pelosi P, Schultz MJ; for the LAS VEGAS; study-investigators; the PROVE Network; and the Clinical Trial Network of the European Society of Anaesthesiology. The effects of preoperative moderate to severe anaemia on length of hospital stay: A propensity score-matched analysis in non-cardiac surgery patients. Eur J Anaesthesiol. 2021 Jun 1;38(6):571-581. doi: 10.1097/EJA.0000000000001412. PMID 33399375
- [Derived] Uhlig C, Neto AS, van der Woude M, Kiss T, Wittenstein J, Shelley B, Scholes H, Hiesmayr M, Vidal Melo MF, Sances D, Coskunfirat N, Pelosi P, Schultz M, Gama de Abreu M; LAS VEGAS# investigators, Protective Ventilation Network (PROVEnet), Clinical Trial Network of the European Society of Anaesthesiology. Intraoperative mechanical ventilation practice in thoracic surgery patients and its association with postoperative pulmonary complications: results of a multicenter prospective observational study. BMC Anesthesiol. 2020 Jul 22;20(1):179. doi: 10.1186/s12871-020-01098-4. PMID 32698775
- [Derived] Cortegiani A, Gregoretti C, Neto AS, Hemmes SNT, Ball L, Canet J, Hiesmayr M, Hollmann MW, Mills GH, Melo MFV, Putensen C, Schmid W, Severgnini P, Wrigge H, Gama de Abreu M, Schultz MJ, Pelosi P; LAS VEGAS Investigators, the PROVE Network, and the Clinical Trial Network of the European Society of Anaesthesiology. Association between night-time surgery and occurrence of intraoperative adverse events and postoperative pulmonary complications. Br J Anaesth. 2019 Mar;122(3):361-369. doi: 10.1016/j.bja.2018.10.063. Epub 2019 Feb 8. PMID 30770054
- [Derived] Ball L, Hemmes SNT, Serpa Neto A, Bluth T, Canet J, Hiesmayr M, Hollmann MW, Mills GH, Vidal Melo MF, Putensen C, Schmid W, Severgnini P, Wrigge H, Gama de Abreu M, Schultz MJ, Pelosi P; LAS VEGAS investigators; PROVE Network; Clinical Trial Network of the European Society of Anaesthesiology. Intraoperative ventilation settings and their associations with postoperative pulmonary complications in obese patients. Br J Anaesth. 2018 Oct;121(4):899-908. doi: 10.1016/j.bja.2018.04.021. Epub 2018 Jun 2. PMID 30236252
- [Derived] Neto AS, da Costa LGV, Hemmes SNT, Canet J, Hedenstierna G, Jaber S, Hiesmayr M, Hollmann MW, Mills GH, Vidal Melo MF, Pearse R, Putensen C, Schmid W, Severgnini P, Wrigge H, Gama de Abreu M, Pelosi P, Schultz MJ; LAS VEGAS. The LAS VEGAS risk score for prediction of postoperative pulmonary complications: An observational study. Eur J Anaesthesiol. 2018 Sep;35(9):691-701. doi: 10.1097/EJA.0000000000000845. PMID 29916860
- [Derived] LAS VEGAS investigators. Epidemiology, practice of ventilation and outcome for patients at increased risk of postoperative pulmonary complications: LAS VEGAS - an observational study in 29 countries. Eur J Anaesthesiol. 2017 Aug;34(8):492-507. doi: 10.1097/EJA.0000000000000646. PMID 28633157
- See also: LAS VEGAS Study Specific Website — https://sites.google.com/site/lasvegasstudy/home